CLINICAL TRIAL: NCT02482896
Title: The Lolland-Falster Health Study
Acronym: LOFUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Region Sjælland (Other)
Collaborators: Lolland Municipality, Denmark (Unknown); Guldborgsund Municipality, Denmark (Unknown)
Responsible Party: Sponsor
Other Study IDs: SJ-421
Record Dates: First submitted 2015-06-01; First posted 2015-06-26 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-06

CONDITIONS: Impaired Health; Disease; Wellbeing; Mental Disorders; Atherosclerosis; Renal Insufficiency, Chronic; Skin Diseases; Urinary Incontinence; Personality; Coronary Disease; Ear Diseases; Nose Diseases; Pharyngeal Diseases; Chronic Disease
MeSH Terms: conditions — Disease; Mental Disorders; Atherosclerosis; Renal Insufficiency, Chronic; Skin Diseases; Urinary Incontinence; Coronary Disease; Ear Diseases; Nose Diseases; Pharyngeal Diseases; Chronic Disease

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, urine, faeces, saliva
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study is a epidemiological, cross-sectional study in a mainly rural area of Denmark in Denmark. Life expectancy is shorter, morbidity is higher, and social problems more prevalent than in the urban areas of the country. The population study aims at examining complexities of environmental, hereditary, lifestyle, and social factors as determinants and predisposing factors for morbidity, health, and quality of life. The study will cover physical, mental, and social dimensions and examine family patterns and subgroups. The study will provide baseline information for later follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Individuals registered in Lolland or Guldborgsund municipality

Exclusion Criteria:

* Adults with incapacity guardianship
* Incapacity to give informed consent
* Individuals with address protection
* Severe physical immobility
* Non-Danish and Non-English speaking

Max Age: 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of Lolland and Guldborgsund municipalities in Denmark.
Sampling Method: Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2016-02; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Health | Cross-sectional, measured once
  Self-administered questionnaires, clinical examination, and biospecimen

SECONDARY OUTCOMES:
Morbidity | Cross-sectional, measured once
  Self-administered questionnaires, clinical examination, and biospecimen
Risk factors | Cross-sectional, measured once
  Self-administered questionnaires, clinical examination, and biospecimen

CONTACTS AND LOCATIONS:
Overall Officials: Knud Rasmussen, Dr. Med., MD, Principal Investigator — Region Sjælland
Locations (1):
- The Lolland-Falster Health Study, Nykøbing Falster, Region Sjælland, Denmark

REFERENCES:
- [Derived] Mortensen SR, Brond JC, Petersen TL, Jepsen R, Dominguez-Navarro F, Skou ST, Grontved A. Association of Device-Measured Habitual Sedentary Activity and Standing Posture With Blood Pressure and Hypertension in Danish Adults: The Lolland-Falster Health Study. J Am Heart Assoc. 2025 Aug 19;14(16):e039133. doi: 10.1161/JAHA.124.039133. Epub 2025 Aug 18. PMID 40820973
- [Derived] Bruun-Rasmussen NE, Napolitano G, Bojesen SE, Ellervik C, Holmager TLF, Rasmussen K, Lynge E. Correlation between allostatic load index and cumulative mortality: a register-based study of Danish municipalities. BMJ Open. 2024 Feb 12;14(2):e075697. doi: 10.1136/bmjopen-2023-075697. PMID 38346879
- [Derived] Mortensen SR, Skou ST, Brond JC, Ried-Larsen M, Petersen TL, Jorgensen LB, Jepsen R, Tang LH, Bruun-Rasmussen NE, Grontved A. Detailed descriptions of physical activity patterns among individuals with diabetes and prediabetes: the Lolland-Falster Health Study. BMJ Open Diabetes Res Care. 2023 Sep;11(5):e003493. doi: 10.1136/bmjdrc-2023-003493. PMID 37699719
- [Derived] Gronlund C, Djurhuus BD, Holm EA, Homoe P. Self-reported dizziness, falls, and self-rated health in a rural population in Denmark. Eur Arch Otorhinolaryngol. 2023 Dec;280(12):5329-5337. doi: 10.1007/s00405-023-08061-2. Epub 2023 Jul 8. PMID 37420013
- [Derived] Sondergaard E, Reventlow S, Siersma V, Nicolaisdottir DR, Jepsen R, Rasmussen K, Moller A. A cross-sectional study of the association between family conflicts and children's health: Lolland-Falster Health Study. Child Care Health Dev. 2023 Nov;49(6):972-984. doi: 10.1111/cch.13108. Epub 2023 Feb 28. PMID 36805605
- [Derived] Petersen TL, Brond JC, Kristensen PL, Aadland E, Grontved A, Jepsen R. Resemblance in Physical Activity in Families with Children in Time Segments during the Week: The Lolland-Falster Health Study. Med Sci Sports Exerc. 2021 Nov 1;53(11):2283-2289. doi: 10.1249/MSS.0000000000002718. PMID 34107506
- [Derived] Jacobsen KK, Jepsen R, Lembeck MA, Nilsson C, Holm E. Associations between the SHARE frailty phenotype and common frailty characteristics: evidence from a large Danish population study. BMJ Open. 2019 Oct 15;9(10):e032597. doi: 10.1136/bmjopen-2019-032597. PMID 31619433
- [Derived] Jepsen R, Egholm CL, Brodersen J, Simonsen E, Grarup J, Cyron A, Ellervik C, Rasmussen K. Lolland-Falster Health Study: Study protocol for a household-based prospective cohort study. Scand J Public Health. 2020 Jun;48(4):382-390. doi: 10.1177/1403494818799613. Epub 2018 Sep 17. PMID 30222051